CLINICAL TRIAL: NCT04043897
Title: Efficacy and Safety of Oral Rifaximin in Patients With Active Microscopic Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eugene F Yen, MD (Other)
Responsible Party: Sponsor-Investigator, Eugene F Yen, MD, Clinical Associate Professor of Medicine, Endeavor Health
Organization: Endeavor Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EH17-360
Record Dates: First submitted 2019-02-14; First posted 2019-08-02 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Microscopic Colitis
Keywords: Microscopic Colitis
MeSH Terms: conditions — Colitis, Microscopic | interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: Patients with a diagnosis of microscopic colitis will receive open-label rifaximin 550mg tid x 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug (Experimental): Patients will receive open-label rifaximin 550mg tid x 4 weeks.
  Interventions: Drug: Rifaximin 550mg

INTERVENTIONS:
Drug: Rifaximin 550mg — Rifaximin 550mg

SUMMARY:
This is an open label study looking at rifaximin therapy for the treatment of microscopic (collagenous or lymphocytic) colitis.

DETAILED DESCRIPTION:
This is an open-label single-arm trial to evaluate the efficacy of Rifaximin in patients with active microscopic colitis (MC). 10 subjects will be asked to take 500mg Rifaximin three times per day for 4 weeks. The primary endpoints will be histologic response and clinical remission (less than 3 stools per day and less than 1 watery stool per day within the prior 7 days. The secondary endpoint will be change of the MC Disease Activity Index (MCDAI).

ELIGIBILITY:
Inclusion Criteria:

* Collagenous colitis (CC) or lymphocytic colitis (LC) diagnosed on colon biopsies reviewed by 2 separate pathologists
* CC will be defined histologically to be the following: thickness of the collagenous subepithelial table >10 micrometer using an ocular micrometer, inflammation in the lamina propria consisting of mainly lymphocytes and plasma cells, lack of crypt architectural distortion, and regenerative-appearing changes in the surface and/or crypt epithelium
* LC will be defined histologically to be the following: intraepithelial lymphocytes >20 per 100 epithelial cells in the subjective area of highest lymphocyte density, inflammation in the lamina propria consisting of mainly lymphocytes and plasma cells, and regenerative-appearing changes in the surface and/or crypt epithelium
* Subjects in active flare, defined as >3 watery/loose stools per day on >4 / 7 days over >4 weeks in the past 3 months.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-29 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of Subject Experiencing Remission of MC Symptoms | 6 weeks
  Remission, which will be define as less than 3 stools per day and less than 1 watery stool per day within the prior 7 days as per Hjortswang criteria, which has been used as the standard definition of remission in most all randomized clinical trials evaluating budesonide and MC. Investigators will also look at number of bowel movements, abdominal pain, incontinence, and nocturnal bowel movements. Symptoms will be compared at Week 0 and Week 6.
Histologic Response for Indications of Disease Severity | 6 weeks
  Our institution has identified histologic parameters associated with more severe disease activity. In collaboration with pathologists, investigators will compare histologic inflammation on patients before and after treatment. Histology will be assessed via standard H&E staining, specifically looking at surface epithelial changes associated with disease severity.

SECONDARY OUTCOMES:
Change of the MC Disease Activity Index (MCDAI) | 6 weeks
  The MCDAI scale was developed to best predict a patient's quality of life as well as approximate a physician's global assessment. In multivariate analysis, the MCDAI demonstrated four independent clinical features associated with the physician global assessment including the number of unformed stools daily, number of nocturnal stools, abdominal pain, and number of episodes of fecal incontinence. These factors were used to develop estimated regression coefficients as weights produced the MCDAI formula: 1.1+0.31 (average number of unformed stools daily over the past week; continuous variable)+0.78 (nocturnal stools over past week, 0=absent, 1=present)+0.22 (maximum abdominal pain over past week, score 1-10)+0.11 (average weight loss per month (lbs))+0.93 (fecal urgency over past week, 0=absent, 1=present)+0.01 (number of episodes of fecal incontinence over past month; continuous variable).
  This will be assessed at Week 0 and at Week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Yen, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No